CLINICAL TRIAL: NCT02154750
Title: Evaluation of AV Delay Optimization vs. Intrinsic Conduction in Patients With Long PR Intervals Receiving Dual Chamber Pacemakers for Symptomatic Bradycardia
Brief Title: AV Delay Optimization vs. Intrinsic Conduction in Pacemaker Patients With Long PR Intervals
Acronym: AV Delay
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Greg Feld, Professor of Medicine, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 130663
Record Dates: First submitted 2014-05-28; First posted 2014-06-03 (Estimated); Results first posted 2025-06-12 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Atrioventricular Block; Sick Sinus Syndrome; Symptomatic Bradycardia; Cardiac Arrhythmia
Keywords: Atrioventricular delay; AV delay; Pacemaker; Sick Sinus Syndrome; Bradycardia; PR interval; Atrioventricular block; AV block; Echocardiography; Arrhythmia; AV optimization
MeSH Terms: conditions — Atrioventricular Block; Sick Sinus Syndrome; Arrhythmias, Cardiac; Bradycardia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Long, fixed AV delay (Active Comparator): Pacemaker will be set to a long, fixed AV delay to minimize ventricular pacing
  Interventions: Device: Long, fixed AV delay
- Short, optimized AV delay (Experimental): Pacemaker will be set to the AV delay that produces the greatest cardiac output in echocardiography for each patient enrolled
  Interventions: Device: Short, optimized AV delay

INTERVENTIONS:
Device: Long, fixed AV delay — Pacemaker will be set to a long, fixed AV delay to minimize ventricular pacing
  Arms: Long, fixed AV delay
Device: Short, optimized AV delay — Pacemaker will be set to the AV delay that produces the greatest cardiac output in echocardiography for each patient enrolled.
  Arms: Short, optimized AV delay

SUMMARY:
This is a randomized, prospective clinical trial to determine the effects of two different pacemaker atrioventricular delay (AV delay) settings on heart function in patients with dual chamber pacemakers implanted for symptomatic bradycardia with long PR intervals (delayed conduction between upper and lower chambers of the heart). The study will compare a long, fixed AV delay (standard) with an optimized AV delay for each individual using echocardiography (experimental).

DETAILED DESCRIPTION:
Cardiac pacing is the only effective treatment for symptomatic sinus node dysfunction. Most patients with preserved left ventricular function receive dual chamber pacemakers; however, right ventricular pacing can have detrimental effects on left ventricular function due to the abnormal electrical and mechanical activation pattern of the ventricles.

Many patients receiving dual chamber pacemakers for symptomatic bradycardia have prolonged intrinsic AV conduction (first degree AV block), and as a result, will receive a significant amount of ventricular pacing if programmed at physiologic AV intervals. As an alternative, many pacemakers can be programmed to minimize ventricular pacing at the expense of allowing longer AV delays. However, these long AV delays may not be physiologic and may also lead to reduced cardiac output. At present the standard of care is either to program the pacemaker at an physiologic "natural" AV delay of about 160 msec or to program the pacemaker with a long AV delay to minimize ventricular pacing.

The main scientific questions being addressed in this study are to evaluate the acute and chronic effects on cardiac output, functional status, sense of well-being, and cardiac remodeling of a long AV delay allowing for intrinsic conduction as compared to an echocardiographically optimized AV delay during dual chamber pacing.

Patients enrolled in the trial will complete a run-in period of two weeks prior to randomization in which pacemakers will be programmed with a long-fixed AV delay to allow intrinsic conduction and minimize ventricular pacing (standard). At two weeks, patients will receive a baseline echocardiogram. To determine optimal AV delay, all patients will undergo echocardiographic analysis at varying AV delays. Optimal AV delay will be defined as the AV delay associated with the largest average aortic Doppler velocity time integral (VTI). Then, patients will be randomized to either the short, optimized (experimental) or long, fixed (standard) AV delay groups. To assess functional status and sense of well-being, patients will complete a six minute walk test and Short Form-36 Medical Outcomes Study Questionnaire. Patients return to clinic for another study visit at 6 months and repeat research procedures, including baseline echocardiogram, questionnaire, and 6 minute walk test.

ELIGIBILITY:
Patient population: Individuals with 1st degree atrioventricular (AV) block who have received a dual chamber pacemaker for symptomatic bradycardia.

Inclusion Criteria:

1. Patients greater than 18 years of age
2. Patients with symptomatic sinus bradycardia
3. Patients who meet standard indications for dual chamber pacemaker implantation
4. Patients who have 1st degree AV block determined by PR interval > 200ms

Exclusion Criteria:

1. Patients with complete or high grade AV block
2. Patients who are unable to complete dual chamber pacemaker implantation for any reason
3. Patients with congestive heart failure determined by a Left Ventricular Ejection Fraction < 45%
4. Patients with persistent atrial fibrillation
5. Sustained premature ventricular contractions (PVCs), premature atrial contractions (PACs), atrial flutter, or other heart conditions that may interfere with echocardiography measurements
6. Patients who are pregnant
7. Patients with Paroxysmal Atrial Fibrillation that have had an episode(s) within 30 days of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2013-06-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory K Feld, MD, Principal Investigator — UCSD Electrophysiology
Locations (1):
- UCSD Sulpizio Cardiovascular Center, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sawhney NS, Waggoner AD, Garhwal S, Chawla MK, Osborn J, Faddis MN. Randomized prospective trial of atrioventricular delay programming for cardiac resynchronization therapy. Heart Rhythm. 2004 Nov;1(5):562-7. doi: 10.1016/j.hrthm.2004.07.006. PMID 15851220
- [Background] Tops LF, Schalij MJ, Bax JJ. The effects of right ventricular apical pacing on ventricular function and dyssynchrony implications for therapy. J Am Coll Cardiol. 2009 Aug 25;54(9):764-76. doi: 10.1016/j.jacc.2009.06.006. PMID 19695453
- [Background] Iliev II, Yamachika S, Muta K, Hayano M, Ishimatsu T, Nakao K, Komiya N, Hirata T, Ueyama C, Yano K. Preserving normal ventricular activation versus atrioventricular delay optimization during pacing: the role of intrinsic atrioventricular conduction and pacing rate. Pacing Clin Electrophysiol. 2000 Jan;23(1):74-83. doi: 10.1111/j.1540-8159.2000.tb00652.x. PMID 10666756
- [Background] Sweeney MO, Ellenbogen KA, Tang AS, Whellan D, Mortensen PT, Giraldi F, Sandler DA, Sherfesee L, Sheldon T; Managed Ventricular Pacing Versus VVI 40 Pacing Trial Investigators. Atrial pacing or ventricular backup-only pacing in implantable cardioverter-defibrillator patients. Heart Rhythm. 2010 Nov;7(11):1552-60. doi: 10.1016/j.hrthm.2010.05.038. Epub 2010 Jun 4. PMID 20685401

RESULTS

PARTICIPANT FLOW:
Groups:
- Long Fixed AV Delay: 12 subjects were enrolled in the long-fixed AV delay group.
- Optimized AV Delay: 11 subjects were enrolled in optimized AV delay group
Period: Overall Study
Arm/Group | Long Fixed AV Delay | Optimized AV Delay
Started | 12 | 11
Completed | 12 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Long, Fixed AV Delay | Short, Optimized AV Delay | Total
Number analyzed (Participants) | 12 | 11 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 11 | 23
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.8 (6.6) | 78.0 (5.7) | 72.7 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 9 | 8 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 11 | 10 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 11 | 23

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Change in Echocardiographic Parameters LV Dimension at End-diastole, LV Dimension at End-systole, and Tricuspid Annular Plane Systolic Excursion (cm) From Baseline to Followup, in Optimized AV Delay Versus Long-fixed AV Delay Groups.
Description: Comparison (∆) of change in echocardiographic parameters left ventricular (LV) dimension at end-diastole, left ventricular (LV) dimension at end-systole, and tricuspid annular plane systolic excursion (cm) from baseline to followup, in Optimized AV delay versus Long-fixed AV delay groups. A reduction LV dimension indicates improvement in function, and an increase in tricuspid annular plane excursion represents an improvement in function.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: cm
Groups:
- Optimized AV Delay: Pacemaker will be set to the AV delay that produces the greatest cardiac output in echocardiography for each patient enrolled
  Short, optimized AV delay: Pacemaker will be set to the AV delay that produces the greatest cardiac output in echocardiography for each patient enrolled.
- Long Fixed AV Delay: Pacemaker will be set to a long, fixed AV delay to minimize ventricular pacing
  Long, fixed AV delay: Pacemaker will be set to a long, fixed AV delay to minimize ventricular pacing
Arm/Group | Optimized AV Delay | Long Fixed AV Delay
Number analyzed (Participants) | 11 | 12
cm
  Left Ventricular Dimension at End-Diastole (LVDd) | -3.1 (6.2) | 0.1 (4.8)
  Left Ventricular Dimension as End-Systole (LVDs) | -4.2 (18.6) | -1.9 (14)
  Tricuspid annular plane systolic excursion | 2.4 (0.5) | 2.3 (0.4)

2. Primary Outcome: Comparison of Echocardiographic Parameters Mitral E Wave Velocity (cm/s) and Mitral A Wave Velocity (cm/s) at Baseline and Followup, in Optimized AV Delay Versus Long-fixed AV Delay Group.
Description: Comparison (∆) of echocardiographic parameters mitral E wave velocity (cm/s) and mitral A wave velocity (cm/s) at baseline and followup, in Optimized AV delay versus Long-fixed AV delay group. An increase in mitral E wave velocity and a decrease in mitral A velocity represent an improvement in function.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: cm/s
Arm/Group | Optimized AV Delay | Long Fixed AV Delay
Number analyzed (Participants) | 11 | 12
cm/s
  ∆ Mitral E wave velocity | -5.5 (16.4) | 0.8 (21.9)
  ∆ Mitral A wave velocity | 3.5 (12.3) | 0.0 (26)

3. Primary Outcome: Comparison of Change in Echocardiographic Parameter ΔE/A and Mean E/e' Ratio (Unitless) From Baseline to Followup, in Optimized AV Delay Versus Long-fixed AV Delay Groups.
Description: Comparison (Δ) of change in echocardiographic parameter ΔE/A and Mean E/e' ratio (unitless) from baseline to followup, in Optimized AV delay versus Long-fixed AV delay groups. An higher delta E/A and mean E/e' ratio represent improvement in function,
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Ratio (unitless)
Arm/Group | Optimized AV Delay | Long Fixed AV Delay
Number analyzed (Participants) | 11 | 12
Ratio (unitless)
  Δ E/A Ratio | 5.8 (32) | -15.9 (31.1)
  Δ Mean E/e' | -1.1 (29.2) | -5.6 (14.4)

4. Primary Outcome: Comparison of Echocardiographic Parameter Deceleration Time (Msec) at Baseline and Followup, in Optimized AV Delay Versus Long-fixed AV Delay Group.
Description: Comparison (∆) of Echocardiographic Parameter Deceleration time (msec) at Baseline and Followup, in Optimized AV Delay Versus Long-fixed AV Delay Group. A reduction in deceleration time represents an improvement in function.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Optimized AV Delay | Long Fixed AV Delay
Number analyzed (Participants) | 11 | 12
msec | 14.6 (15.7) | 2.1 (20.2)

5. Primary Outcome: Comparison of Change in Echocardiographic Parameters LVED End Diastolic Volume Index, LVES Volume Index, Maximum LA Volume Index, and Minimum LA Volume Index (ml/m2) From Baseline to Follow-up, in Optimized AV Delay Versus Long-fixed AV Delay Groups.
Description: Comparison of change in echocardiographic parameters left ventricular end diastolic (LVED) volume index, left ventricular end systolic (LVES) volume index, maximum left atrial (LA) volume index, and minimum left atrial (LA) volume index (ml/m2) from baseline to follow-up, in Optimized AV delay versus Long-fixed AV delay groups. A reduction in volume indexes represents an improvement in function.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: ml/m2
Arm/Group | Optimized AV Delay | Long Fixed AV Delay
Number analyzed (Participants) | 11 | 12
ml/m2
  Left ventricular end diastolic volume index | -13.2 (11) | 5.8 (18.7)
  Left ventricular end systolic volume index | -16.4 (13.6) | 6.7 (22.9)
  Maximum left atrial volume index | -9.7 (40.9) | 0.6 (25.4)
  Minimum left atrial volume index | -9.1 (42.1) | 1.8 (28.6)

6. Primary Outcome: Comparison of Change in Echocardiographic Parameters Left Ventricular Ejection Fraction and Global Longitudinal Strain (%) From Baseline to Followup, in Optimized AV Delay Versus Long-fixed AV Delay Groups.
Description: Comparison (∆) of Change in Echocardiographic Parameters Left Ventricular Ejection Fraction and Global Longitudinal Strain (%) From Baseline to Followup, in Optimized AV Delay Versus Long-fixed AV Delay Groups. An increase in left ventricular ejection time represents an improvement in function. A more negative global longitudinal strain % represents an improvement in function.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Optimized AV Delay | Long Fixed AV Delay
Number analyzed (Participants) | 11 | 12
percentage
  Left Ventricular Ejection Fraction | 4.4 (13.1) | -0.7 (8.7)
  Global Longitudinal Strain | 5.5 (16.1) | -11.8 (17.8)

7. Primary Outcome: Comparison of Change in Echocardiographic Parameters Tricuspid Regurgitation (TR) Velocity m/s From Baseline to Followup, in Optimized AV Delay Versus Long-fixed AV Delay Groups.
Description: Comparison (∆) of Change in Echocardiographic Parameters Tricuspid Regurgitation (TR) velocity m/s From Baseline to Followup, in Optimized AV Delay Versus Long-fixed AV Delay Groups. An reduction in tricuspid regurgitation velocity represents an improvement in function.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: m/sec
Arm/Group | Optimized AV Delay | Long Fixed AV Delay
Number analyzed (Participants) | 11 | 12
m/sec | 2.2 (0.3) | 2.2 (0.5)

8. Primary Outcome: Comparison of Change in Echocardiographic Parameters Left Ventricular Mass (gm) From Baseline to Followup, in Optimized AV Delay Versus Long-fixed AV Delay Groups.
Description: Comparison (∆) of Change in Echocardiographic Parameters left ventricular mass (gm) From Baseline to Followup, in Optimized AV Delay Versus Long-fixed AV Delay Groups. A reduction in left ventricular mass represents an improvement in function.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: gm
Arm/Group | Optimized AV Delay | Long Fixed AV Delay
Number analyzed (Participants) | 11 | 12
gm | 142.8 (21) | 148.4 (23.2)

9. Secondary Outcome: Comparison of Measured Distance Walked in 6 Minutes in Meters From Baseline and Followup, in Optimized AV Delay Group Versus Long-fixed AV Delay Group.
Description: Comparison (∆) of measured distance walked in 6 minutes in meters from baseline and followup, in Optimized AV delay group versus Long-fixed AV delay group. An increase in distance walked during the 6 minute walk test represents an improvement in function.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: meters
Groups:
- Long-fixed AV Delay: Pacemaker will be set to a long, fixed AV delay to minimize ventricular pacing
  Long, fixed AV delay: Pacemaker will be set to a long, fixed AV delay to minimize ventricular pacing
Arm/Group | Optimized AV Delay | Long-fixed AV Delay
Number analyzed (Participants) | 11 | 12
meters | 368.7 (71.8) | 473.8 (83.2)

ADVERSE EVENTS:
Time Frame: 6 years
Groups:
- Intervention - Long Fixed AV Delay: 12 subjects were enrolled in the long fixed AV delay group.
- Intervention - Optimized AV Delay: 11 subjects were enrolled in the optimized AV delay group.
Arm/Group | Intervention - Long Fixed AV Delay | Intervention - Optimized AV Delay
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/11
Other Adverse Events (participants affected / at risk) | 0/12 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-11-15): https://cdn.clinicaltrials.gov/large-docs/50/NCT02154750/Prot_000.pdf
  • Statistical Analysis Plan (2024-11-15): https://cdn.clinicaltrials.gov/large-docs/50/NCT02154750/SAP_001.pdf